CLINICAL TRIAL: NCT02045706
Title: A Randomized Prospective Trial to Measure Health-Related Behavioral Changes in Local Villagers Following The Implementation of a Village Health Team Program Facilitated by The Ugandan Ministry of Health and US Health Volunteers
Brief Title: The Impact of Community Health Worker Training by US Health Volunteers on the Health of Rural Ugandans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward O'Neil Jr, M.D. (Other)
Collaborators: Washington University School of Medicine (Other); Makerere University (Other); Peace Corps (Other); Uganda Chartered Health Net (Unknown); University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor-Investigator, Edward O'Neil Jr, M.D., President of Omni Med, Omni Med
Organization: Omni Med (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SS 2486; #81090 (Other Grant/Funding Number: Award # 81090, Tufts University Charlton Grant)
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Community Health Workers; Service; Volunteerism; Health Behaviors
MeSH Terms: conditions — Behavior; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community Health Worker Trainings (Experimental): Trained community health workers (CHW) (one per 25 households), conducted a focus group and four quarterly meetings. CHWs were then responsible for 25 households where they would teach preventive health, track health data for the Ministry, and refer sick cases (700 households total). Staff and volunteers also conducted home visits and handed out printed summaries. We also worked with the local villagers and community health workers to construct 3 protected water sources in the Intervention areas.
  Interventions: Other: Community Health Worker Trainings
- Control Group (No Intervention): The Control Group was comprised of similar households to the Intervention Group (n = 700). In these villages, however, we did not instill the community health worker program until after the trial was completed.

INTERVENTIONS:
Other: Community Health Worker Trainings
  Other Names: United States Peace Corps; Uganda Ministry of Health; Village Health Teams
  Arms: Community Health Worker Trainings

SUMMARY:
There are many trials measuring the impact of service work on volunteers themselves, but few studies measuring the impact of service on the local people. The purpose of this trial is to determine whether US and Ugandan health volunteers can make a measurable impact on the health of rural Ugandan villagers.

DETAILED DESCRIPTION:
The goal of this research is to measure a change in the behaviors of local villagers in the Mukono District (just east of Kampala, Uganda) following the implementation of the Ministry of Health's Village Health Team Program facilitated by US Health Volunteers. Our NGO (non-governmental organization), Omni Med, has partnered with the Ministry of Health in Kampala and Mukono to facilitate its Village Health Team (VHT) program. Our volunteers facilitate training of VHTs and then conduct follow up home visits with these VHTs. During the trainings and follow up visits we stress the health practices in the Ministry's training program that have been shown to make the biggest impact on local health such as: exclusive breast-feeding for 9 months, use of oral rehydration therapy (ORT), antibiotics for pneumonia, timely antimalarial use, use of insecticide treated nets (ITNs), clean water, improved sanitation, Vitamin A supplementation and vaccination, antenatal visits and tetanus immunization for pregnant women, etc. Our pre-trial assumption is that local villagers will use this knowledge to improve their own health; and that the VHTs are the ideal messengers to deliver this knowledge. While the Ministry has trained over 83,000 VHTs nationally, there are no objective studies measuring impact on host communities. This will be the first and could prove an important means to promote the program nationally and internationally.

The primary objective of this research is to measure the efficacy of the VHT program in Uganda. While this program has become a priority of the Ministry of Health, there is to date no clear randomized, prospective trial measuring its impact. This will thus fill a current gap using data obtained from 1190 households. A second objective is to demonstrate measurable results of a global service program. There is very little impact data despite huge interest in service from many in the world's wealthiest countries. A third objective is to provide an objective measure of efficacy to the United States Peace Corps, which despite 50 years of activities, has little data demonstrating its true value; several Peace Corps Volunteers are working in this program in Mukono.

ELIGIBILITY:
Inclusion Criteria: Household with children under age five -

Exclusion Criteria: No children under age five in the household

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1419 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Questionnaire on health behaviors before and after implementation of a community health worker program | One year
  A detailed questionnaire about local health behaviors was employed by Uganda Chartered Health Net in villages randomized to control and intervention areas in two parishes in rural Uganda. Data was collected in both areas before and after implementation of a Ministry of Health mandated community health worker program over a one year period. Key outcome measures were then plugged into the Lives Saved Tool (LIST) to determine changes in infant and under-5 mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Edward J O'Neil Jr, MD, Principal Investigator — Omni Med
Locations (2):
- Omni Med, Newton, Massachusetts, United States
- Uganda Chartered Health Net, Kampala, Uganda